CLINICAL TRIAL: NCT05027815
Title: A Phase 1/2a Study of Cryopreserved Ex Vivo Expanded Polyclonal CD4+CD127lo/-CD25+ T Regulatory Cells (cePolyTregs) for the Treatment of Acute Respiratory Distress Syndrome (ARDS) Associated With SARS-CoV-2 Infection (regARDS)
Brief Title: Tregs for the Treatment of Acute Respiratory Distress Syndrome (ARDS) Associated With COVID-19 (regARDS)
Acronym: regARDS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decrease in COVID-19 cases made further enrollment infeasible.
Sponsor: Jeffrey Bluestone (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor-Investigator, Jeffrey Bluestone, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UCSF-cePolyTregs-01; 3UM1AI109565-08S3 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2021-08-30 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Acute Respiratory Distress Syndrome Due to Disease Caused by 2019-nCoV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- cePolyTregs 100 x10^6 cells Open Label (Experimental): single dose of 100 x 10^6 cells by IV infusion
  Interventions: Biological: Cryopreserved Ex Vivo Expanded Polyclonal CD4+CD127lo/-CD25+ T Regulatory Cells
- cePolyTregs 200 x10^6 cells Open Label (Experimental): single dose of 200 x 10^6 cells by IV infusion
  Interventions: Biological: Cryopreserved Ex Vivo Expanded Polyclonal CD4+CD127lo/-CD25+ T Regulatory Cells
- cePolyTregs 400 x10^6 cells Open Label (Experimental): single dose of 400 x 10^6 cells by IV infusion
  Interventions: Biological: Cryopreserved Ex Vivo Expanded Polyclonal CD4+CD127lo/-CD25+ T Regulatory Cells

INTERVENTIONS:
Biological: Cryopreserved Ex Vivo Expanded Polyclonal CD4+CD127lo/-CD25+ T Regulatory Cells — cryopreserved cellular therapy product in cryostor CS5, for IV infusion
  Other Names: cePolyTregs

SUMMARY:
In patients with Acute Respiratory Distress Syndrome (ARDS) associated with COVID-19 inflammatory syndrome, the administration of Treg cells is a novel treatment complementary to other pharmacologic interventions that potentially can reduce lung inflammation, promote lung tissue repair, and significantly improve clinical outcomes. This trial is to evaluate the impact of a single IV dose of cePolyTregs given to ARDS patients with COVID-19 inflammatory syndrome.

DETAILED DESCRIPTION:
Tregs are a subset of CD4+ T cells that function to maintain immune system balance. The function of Tregs in maintaining immune tolerance can be harnessed through Treg cell therapy for treating various immunological diseases. Adoptive Tregs therapies have been shown to be effective in dozens of animal models, including models of virus-induced ARDS. This is a Phase 1 study to evaluate the safety and tolerability of cePolyTregs in subjects with ARDS associated with SARS-CoV-2 infection. The study is an open-label Phase 1 study to assess escalating doses of cePolyTregs administered as a single IV dose. The study will include up to 3 cohorts of 3 to 6 subjects/cohort followed for a total of 12 weeks. All subjects will receive standard of care treatment for COVID-19, including dexamethasone per institutional guidelines and other approved therapies for ARDS associated with SARS-CoV-2 infection per institutional guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ARDS and respiratory failure requiring mechanical ventilation for less than 72 hours at the time of enrollment
* PaO2/FiO2 < 300 and PEEP > 5
* Male or female, age 18 to 70 years at Screening
* Weight > 40 kg
* Documented diagnosis of infection with SARS-CoV-2 virus by PCR
* Chest imaging (radiograph or CT scan) with abnormalities consistent with COVID-19 pneumonia that could not be explained by effusions, pulmonary collapse, or nodules; and respiratory failure that could not be explained by cardiac failure or fluid overload
* Females of childbearing potential and males must use effective contraception practices from Screening until 28 days after the EOS visit
* Females of childbearing potential must have a negative pregnancy test at Screening and within 24 hours prior to dosing of study drug
* Able to provide Informed Consent, either by self or by medical proxy
* Willing and able to comply with this protocol for the entire duration of the study

Exclusion Criteria:

* Any history or sign of significant chronic active or recurrent infection or screening laboratory evidence consistent with a significant chronic active or recurrent infection requiring treatment with antibiotics, antivirals or antifungals (other than SARS-CoV-2); ongoing antimicrobial treatments will not be exclusionary if, in the opinion of the investigator, no active infection is present (other than SARS-CoV-2)
* Receiving extracorporeal membrane oxygenation therapy
* Moribund patients not expected to survive 24 hours after enrollment based on clinical assessment
* History of significant underlying pulmonary disease (requiring home oxygen), renal disease (requiring dialysis for chronic kidney disease), hepatic disease (Child-Pugh score ≥ 7), or known history of cirrhosis.
* Known or suspected immunodeficiency disease
* Positive serology for HBV, HCV, or HIV at Screening
* Abnormal CBC defined by:

  * Platelet count < 75,000/mm3
  * White blood cell count < 2500/mm3
  * Absolute neutrophil count < 500/mm3
* History of bone marrow or stem cell transplantation
* Received any type of live attenuated vaccine < 1 month prior to Screening or is planning to receive any such live attenuated vaccine over the course of the study
* History of lung cancer or any other malignancy requiring active treatment, except adequately treated basal cell carcinoma or in situ carcinoma of the uterine cervix
* Any female who is pregnant or breastfeeding, or any female who is planning to become pregnant during the study and follow-up period
* Any condition that, in the investigator's opinion, may compromise study participation, present a safety risk to the subject, or may confound the interpretation of the study results
* A QT duration corrected for heart rate by Fridericia's formula (QTcF) > 450 millisecond (msec) for males or > 470 msec for females, based on either single or averaged QTcF values of triplicate ECGs obtained over a 3-minute interval
* Currently enrolled in another investigational device or drug study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maor Sauler, MD, Study Chair — Yale University
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from participating medical centers with the first participant consented September 23, 2021 and the last participant consented February 10, 2022.
Pre-assignment Details: Of 7 participants consented, 4 met eligibility criteria and were assigned to a treatment arm. Three were enrolled in the 100x10^6 cells arm, and one was enrolled in the 200 x 10^6 cells arm.
Period: Overall Study
Arm/Group | cePolyTregs 100 x10^6 Cells Open Label | cePolyTregs 200 x10^6 Cells Open Label
Started | 3 | 1
Completed | 1 | 0
Not Completed | 2 | 1
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | cePolyTregs 100 x10^6 Cells Open Label | cePolyTregs 200 x10^6 Cells Open Label | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLT is defined as any related treatment-emergent adverse event (TEAE) with a National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE 5.0) grade ≥ 3 which also represents a shift from baseline clinical status of ≥ 1 NCI CTCAE grade
Time Frame: 28 days post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | cePolyTregs 100 x10^6 Cells Open Label | cePolyTregs 200 x10^6 Cells Open Label
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 84 days post treatment
Arm/Group | cePolyTregs 100 x10^6 Cells Open Label | cePolyTregs 200 x10^6 Cells Open Label
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/1
Other Adverse Events (participants affected / at risk) | 2/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cePolyTregs 100 x10^6 Cells Open Label (N=3) | cePolyTregs 200 x10^6 Cells Open Label (N=1)
Renal Failure requiring renal replacement therapy by CRRT (Renal and urinary disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Refractory Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ventilator-Associated Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cePolyTregs 100 x10^6 Cells Open Label (N=3) | cePolyTregs 200 x10^6 Cells Open Label (N=1)
Pneumonmediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated early due to a decline in the available participants, which prevent the analysis of some secondary and exploratory endpoints from completion as initially planned. The safety and tolerability, and recommended phase 2 dose can not be determined based on the limited data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT05027815/Prot_SAP_000.pdf